CLINICAL TRIAL: NCT05984745
Title: Effect of Coenzyme Q10 on the Outcome of Metabolic Dysfunction-Associated Fatty Liver Disease Patients
Brief Title: Effect of CoQ10 on the Outcome of MAFLD Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Talaat, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CoQ10 in MAFLD Patients
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Fatty Liver; NAFLD
Keywords: Coenzyme Q10; Liver steatosis; TNF alpha; Fatty Liver; Inflammation; MAFLD; CoQ10; Ubiquinone; Liver Disease
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease; Inflammation; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Patients will receive the standard conventional care which is mainly therapeutic life changes
- Test Group (Experimental): Patients will receive Coenzyme Q10 Forte® (MEPACO Pharmaceutical Company, Cairo, Egypt) capsules in a dose of 100 mg twice per day 1 capsule every 12 hours for twelve weeks, in addition to the standard conventional care.
  Interventions: Drug: Coenzyme Q10 Forte® capsules

INTERVENTIONS:
Drug: Coenzyme Q10 Forte® capsules — Coenzyme Q10 in the form of soft gelatin capsules, each capsule containing 100 mg
  Arms: Test Group

SUMMARY:
So far there has been no universal treatment for MAFLD since it has a complex etiology that involves ethnic, genetic, metabolic and environmental factors. However, therapeutic life changes including: diet, weight loss, and physical activity remain the cornerstone of treatment and is recommended by both American and European associations.

Inflammatory biomarkers, such as tumor necrosis factor-alpha, and adipokines play key roles in the pathogenesis of MAFLD, hence, the anti-inflammatory and antioxidant effects of coenzyme Q10 especially at high doses that have not been tested are hypothesized to have a beneficial role in improving the systemic inflammation and biochemical variables.

This study is conducted to test this hypothesis

DETAILED DESCRIPTION:
The liver disease with the most continuously rising prevalence rates is metabolic-dysfunction associated fatty liver disease (MAFLD), making us arrive at a conclusion that it might be the liver disease epidemic of the 21st century. It is increasingly diagnosed in many developed and developing countries and is considered the most common cause of chronic liver disease among patients with type 2 diabetes mellitus (T2DM). By 2030, it will be the leading cause for hepatocellular carcinoma (HCC) related liver transplantation (LTx) in western countries.

A number of studies have suggested that metabolic associated co-morbidities, such as obesity, type 2 DM, CVD, dyslipidemia, hypertension, metabolic syndrome, hypothyroidism, OSAS, PCOS are major risk factors for MAFLD.

It encompasses a wide spectrum of histological pattern, ranging from simple steatosis to steatohepatitis, fibrosis and cirrhosis.

The global prevalence of MAFLD is currently estimated to be 25%, but the highest rates are reported from the Middle East 31.8% and South America 30.5%, followed by Asia 27.4%, the USA 24% and Europe 23.7%, whereas MAFLD is less common in Africa 13.5%.

Coenzyme Q10 (CoQ10) or ubiquinone is a lipid-soluble and vitamin-like compound, which acts as a pivotal cofactor in the mitochondrial respiratory chain in addition to its role as a natural scavenger of free radicals. It is synthesized by cells of the body and also found in abundance in the human diet. Recent evidence suggests that CoQ10 supplementation might be useful in improving and preventing pathological conditions such as metabolic syndrome, hypertension, diabetes, liver diseases, and insulin resistance Because of its antioxidant activity, it seems that CoQ10 can prevent activation of the inflammatory signaling pathway. Many studies have shown that administration of CoQ10 reduced hepatic oxidative stress and inflammation. Also, other studies observed that CoQ10 supplementation reduced TNF-α production and serum levels of liver aminotransferase and decreased NF-kB expression. In addition, a previously published study showed that a dose of 100 mg/day of CoQ10 for 4 weeks can improve serum AST levels, total antioxidant capacity and waist circumference, but it had a non-significant effect on insulin resistance and MDA levels. The same result was found in the study by Esfahani et al. reporting improvement in AST and ALT concentrations and lower grades of portal inflammation and hepatocellular liver necrosis in thioacetamide-induced liver damage in rats. Yet, some contradicting results were reported by Hodgson et al. were they found a non-significant reduction in body weight after CoQ10 supplementation in patients with T2DM. These contradictions were addressed by Faresi et al. where they tested the effect of the same oral dose of CoQ10 used by Farhangi et al. for 12 weeks, where it had beneficial effects on serum levels of TNF-a, hs-CRP, hepatic enzymes, adiponectin, and NAFLD grades as well as near-significant changes in serum leptin among patients with NAFLD. However, serum IL-6 levels and AAR remained unchanged after CoQ10 supplementation.

Till this day, only a few small studies tried to investigate the effect of CoQ10 administration on the degree of steatosis in MAFLD patients and their results failed to show a clear effect, due to the conflicting and limited data. Hence, this encouraged us to study the efficacy and tolerability of a higher dose of CoQ10 especially that it can be safely administered up to a dose of 1200 mg/day. In addition, CoQ10 showed promising effects in previous studies, so the general recommendation was to study its effect in a larger study population, for longer periods.

ELIGIBILITY:
Inclusion Criteria:

All study subjects and prior to consenting to the ICF, laboratory and imaging work-up will be evaluated for the presence of three out of five criteria for metabolic dysregulation in the context of metabolic -dysfunction associated fatty liver disease (MAFLD):

1. Waist circumference (WC) ≥ 102/88 cm for men and women respectively.
2. HDL cholesterol <40 mg/dl in men and <50 mg/dl in women or on specific drug therapy.
3. Plasma Triglycerides ≥ 150 mg/dl or on specific drug therapy.
4. Blood pressure ≥130 and/or ≥ 85 or on specific anti-hypertensive therapy.
5. Fasting blood glucose ≥ 100 mg/dl or on specific anti hyperglycemic therapy

   * Patients who agree to sign an informed consent
   * Adult patients >18 years old.
   * Males and females
   * Willing to comply with procedures and follow up
   * Elevated serum transaminases (1-4 times the ULN)
   * Imaging evidence of fatty liver:

pelviabdominal ultrasound and Fibro- CAP study

Exclusion Criteria:

* Pregnancy or lactating
* Physical or mental abnormalities
* HCV infection
* HBV infection
* Anaemia
* Thrombocytopenia
* Haematological malignancies
* Ongoing alcoholism (Male: >30g/day, Female: >20g/day)
* Patients with renal failure
* Autoimmune hepatitis
* Celiac disease
* Wilson's disease
* Hemochromatosis
* Drugs: Tamoxifen, Valproic acid, Amiodarone, Methotrexate, Steroids, Anticoagulants, All anti-oxidative stress agents, Cos, IUD
* Chronic use of systematically immunosuppressive agent or drugs that can affect liver profile.
* Hypo/Hyper-thyroidism
* Bypass surgeries
* TPN (Total Parenteral Nutrition)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in liver steatosis degree | Baseline and at 12 weeks
  Improvement in steatosis degree will be assessed using Fibro-CAP scoring measured in decibels per meter (dB/m) and ranges from 100-400, where 238 to 260 dB/m represents 11-33% fatty change in the liver, 260 to 290 dB/m represents 34-66% fatty change in the liver and > 290 dB/m represents almost 67% or more fatty change in the liver.

SECONDARY OUTCOMES:
Change in serum levels of tumor necrosis factor-alpha (TNF-α) 3 months post treatment with Coenzyme Q10 | Baseline and at 12 weeks
  TNF-α levels will be assessed in serum
Change in serum levels of cytokeratin-18 (CK-18) 3 months post treatment with Coenzyme Q10 | Baseline and at 12 weeks
  CK-18 levels will be assessed in serum
Change in serum levels of liver transaminases (AST and ALT) 3 months post treatment with Coenzyme Q10 | Baseline and at 12 weeks
  Levels of alanine transaminase (ALT) and aspartate aminotransferase (AST) will be measured in serum where normal serum ALT is 7-56 U/L and normal serum AST is 0 to 35 U/L.
Study the drug's effect on kidney functions by measuring serum creatinine levels | Baseline and at 12 weeks
  Serum creatinine levels will be measured where the normal range is 0.74 to 1.35 mg/dL (61.9 to 114.9 µmol/L) for men and 0.59 to 1.04 mg/dL (53 to 97.2 µmol/L) for women
Change in the quality of life of MAFLD patients | Baseline and at 12 weeks
  Quality of life will be assessed using the Chronic Liver Disease (CLD) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- National Hepatology and tropical medicine research institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] McPherson S, Hardy T, Henderson E, Burt AD, Day CP, Anstee QM. Evidence of NAFLD progression from steatosis to fibrosing-steatohepatitis using paired biopsies: implications for prognosis and clinical management. J Hepatol. 2015 May;62(5):1148-55. doi: 10.1016/j.jhep.2014.11.034. Epub 2014 Dec 1. PMID 25477264
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Alam MA, Rahman MM. Mitochondrial dysfunction in obesity: potential benefit and mechanism of Co-enzyme Q10 supplementation in metabolic syndrome. J Diabetes Metab Disord. 2014 May 23;13:60. doi: 10.1186/2251-6581-13-60. eCollection 2014. PMID 24932457
- [Background] Fuller B, Smith D, Howerton A, Kern D. Anti-inflammatory effects of CoQ10 and colorless carotenoids. J Cosmet Dermatol. 2006 Mar;5(1):30-8. doi: 10.1111/j.1473-2165.2006.00220.x. PMID 17173569
- [Background] Sohet FM, Neyrinck AM, Pachikian BD, de Backer FC, Bindels LB, Niklowitz P, Menke T, Cani PD, Delzenne NM. Coenzyme Q10 supplementation lowers hepatic oxidative stress and inflammation associated with diet-induced obesity in mice. Biochem Pharmacol. 2009 Dec 1;78(11):1391-400. doi: 10.1016/j.bcp.2009.07.008. Epub 2009 Jul 23. PMID 19632207
- [Background] Bravo E, Palleschi S, Rossi B, Napolitano M, Tiano L, D'Amore E, Botham KM. Coenzyme Q metabolism is disturbed in high fat diet-induced non-alcoholic fatty liver disease in rats. Int J Mol Sci. 2012;13(2):1644-1657. doi: 10.3390/ijms13021644. Epub 2012 Feb 2. PMID 22408414
- [Background] Ashkani Esfahani S, Esmaeilzadeh E, Bagheri F, Emami Y, Farjam M. The effect of co-enzyme q10 on acute liver damage in rats, a biochemical and pathological study. Hepat Mon. 2013 Aug 27;13(8):e13685. doi: 10.5812/hepatmon.13685. eCollection 2013. No abstract available. PMID 24130601
- [Background] Farsi F, Mohammadshahi M, Alavinejad P, Rezazadeh A, Zarei M, Engali KA. Functions of Coenzyme Q10 Supplementation on Liver Enzymes, Markers of Systemic Inflammation, and Adipokines in Patients Affected by Nonalcoholic Fatty Liver Disease: A Double-Blind, Placebo-Controlled, Randomized Clinical Trial. J Am Coll Nutr. 2016 May-Jun;35(4):346-53. doi: 10.1080/07315724.2015.1021057. Epub 2015 Jul 9. PMID 26156412
- [Background] Vrentzos E, Ikonomidis I, Pavlidis G, Katogiannis K, Korakas E, Kountouri A, Pliouta L, Michalopoulou E, Pelekanou E, Boumpas D, Lambadiari V. Six-month supplementation with high dose coenzyme Q10 improves liver steatosis, endothelial, vascular and myocardial function in patients with metabolic-dysfunction associated steatotic liver disease: a randomized double-blind, placebo-controlled trial. Cardiovasc Diabetol. 2024 Jul 10;23(1):245. doi: 10.1186/s12933-024-02326-8. PMID 38987784
- [Background] Allen AM, Therneau TM, Larson JJ, Coward A, Somers VK, Kamath PS. Nonalcoholic fatty liver disease incidence and impact on metabolic burden and death: A 20 year-community study. Hepatology. 2018 May;67(5):1726-1736. doi: 10.1002/hep.29546. Epub 2018 Mar 23. PMID 28941364